CLINICAL TRIAL: NCT00906126
Title: Oral Misoprostol for Labor Augmentation: A Dose-Finding Pilot Study
Brief Title: Oral Misoprostol for Labor Augmentation: A Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Kathryn Villano, M.D., University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 122006051
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Arrest of Dilation in Labor
Keywords: oral misoprostol; labor augmentation; arrest of dilation; nulliparous
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Oral Misoprostol 1 (Experimental): Oral misoprostol 25 micrograms every 4 hours for up to two doses.
  Interventions: Drug: Misoprostol
- Oral Misoprostol 2 (Experimental): Oral misoprostol 50 micrograms every 4 hours for up to two doses.
  Interventions: Drug: Misoprostol
- Oral Misoprostol 3 (Experimental): Oral misoprostol 100 micrograms every 4 hours for up to two doses.
  Interventions: Drug: Misoprostol
- Oral Misoprostol 4 (Experimental): Oral Misoprostol 50 micrograms every 2 hours for up to two doses.
  Interventions: Drug: Misoprostol
- Oral Misoprostol 5 (Experimental): Oral Misoprostol 75 micrograms every 4 hours for up to two doses.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Oral misoprostol
  Other Names: Cytotec

SUMMARY:
A phase I, open-label trial to determine a safe dose of oral misoprostol required to augment labor in nulliparous women diagnosed with arrest of dilation.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous
* gestational age of at least 36 weeks
* singleton gestation
* cephalic presentation
* reassuring fetal heart rate
* 4 cm or greater cervical dilation
* ruptured membranes with clear amnionic fluid
* intrauterine pressure catheter in place
* less than 200 MVU's

Exclusion Criteria:

* non-reassuring fetal heart rate
* meconium-stained amnionic fluid
* previous uterine incision
* maternal fever
* pregnancy-induced hypertension or other pregnancy-related complications
* known fetal anomalies
* placenta previa or unexplained vaginal bleeding
* estimated fetal weight of 4,500 grams or greater
* evidence of cephalopelvic disproportion
* any moderate or severe preexisting disease
* contraindication to the use of prostaglandins

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2007-04; Primary Completion 2008-09 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
uterine hyperstimulation

SECONDARY OUTCOMES:
adequate uterine activity
need for oxytocin augmentation
time from administration of study drug to delivery
route of delivery and indications
maternal and neonatal infectious morbidity
neonatal outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn S Villano, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States